CLINICAL TRIAL: NCT02885701
Title: A Prospective, Randomized Controlled Study of Splinting After Mini-Open Carpal Tunnel Release
Brief Title: Splinting After Mini-Open Carpal Tunnel Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anthony L. Logli (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor-Investigator, Anthony L. Logli, Student Doctor, OrthoIllinois
Organization: OrthoIllinois (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWA00009558
Record Dates: First submitted 2016-08-22; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: postoperative dressing; postoperative splint; mini-open carpal tunnel release
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- No splint (Experimental)
  Interventions: Other: No Splint
- Removable Splint (Experimental)
  Interventions: Other: Removable Splint
- Non-removable Splint (Experimental)
  Interventions: Other: Non-removable Splint

INTERVENTIONS:
Other: No Splint — The no splint group received a soft dressing consisting of an occlusive petroleum gauze strip (Xeroform, Mansfield, MA) over the wound, one folded 4x4 gauze, and a single wrap of roll gauze around the hand, and the wrist was placed and secured by a Coban wrap (3M, St. Paul, MN). The dressing permitted wrist and finger motion. Patients were further instructed to remove the dressing at five days and place an adhesive bandage (Band-Aid, Johnson & Johnson, New Brunswick, NJ) over the incision.
  Arms: No splint
Other: Removable Splint — The removable splint group received a V-strap Wrist support (Medical Specialties, Inc., Charlotte, NC) placed over the identical soft dressing that was placed on the no splint group. The cock-up wrist splint was designed to keep the wrist fixed in a 20 degree extended wrist position. Patients were instructed to wear the splint for comfort as needed during day and night. While the patient was wearing the cock-up splint, only finger motion was permitted. Wrist motion was permitted when the cock-up splint was removed.
  Arms: Removable Splint
Other: Non-removable Splint — The plaster non-removable splint group received an occlusive petroleum gauze strip placed over the wound, followed by a 4X4 gauze, and a Webril cotton roll wrap (Covidien, Inc., Covidien, Ireland). A 4- inch, 15-layer thick plaster splint was placed across the volar wrist and molded to keep the wrist in approximately 20 degrees of extension allowing full digital range of motion (ROM). The splint was to be kept dry and not removed by the patient.
  Arms: Non-removable Splint

SUMMARY:
The purpose of this study is to determine if any difference exists among 3 different postoperative splinting regimens- no splint, removable splint, and plaster non-removable splint- following mini-open carpal tunnel release (CTR) surgery.

DETAILED DESCRIPTION:
We sought to determine if any significant difference in patient-reported or clinical outcomes existed among 3 different postoperative splinting regimens- no splint, removable splint, and plaster non-removable splint- following mini-open carpal tunnel release (CTR) surgery for symptomatic, isolated, nerve conduction study positive carpal tunnel syndrome (CTS).

A total of 249 patients received a mini-open CTR and were subsequently randomized into 1 of the 3 splinting regimens to be removed at the first postoperative visit 10-14 days later. Patient-reported outcomes included QuickDASH surveys, Levine-Katz Symptom Severity Scale (SSS) and Functional Status Scale (FSS) and Pain at Rest and in Action using a Numerical Pain Rating Scale (NPRS). Clinical outcomes included wrist range of motion (ROM), grip and lateral pinch strengths. All outcomes were evaluated bilaterally at 10-14 days, 6 weeks, 3 months, 6 months and 12 months after surgery. Demographic information was obtained preoperatively and complications were observed for and recorded throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Patients were required to have failed conservative treatment for symptomatic, isolated, nerve conduction study positive CTS.

Exclusion Criteria:

* Exclusion criteria omitted patients who presented with acute onset CTS, concomitant peripheral neuropathy, metabolic disease, postoperative recurring CTS, or who required another operative procedure during carpal tunnel release.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2010-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
QuickDASH | 10-14 days postoperatively
  The Quick Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure was designed in 1998 with the goal of providing a more accurate depiction of the everyday symptoms and handicaps exclusively experienced by a patient with an upper extremity musculoskeletal condition. Designed as a patient-completed questionnaire, the DASH Outcome Measure can be administered multiple times throughout patient care to measure changes in function and symptoms over time
Levine-Katz Symptom Severity Scale (SSS) | 10-14 days postoperatively
  The Levine-Katz Symptom Severity Scale (SSS) assesses pain, weakness, and sensation with 11 questions the patient rates on a 5-point scale with 5 indicating the most difficult; the average score is reported.
Numerical Pain Rating Scale | 10-14 days postoperatively
  Patients are asked to describe their level of pain intensity over the last 24 hours. The pain scale anchor points 0 and 10 correspond to no pain and worst imaginable pain, respectively. The NPRS can be used multiple times throughout patient care, but has the greatest value in describing post-operative pain-related morbidity.
Grip Strength | 10-14 days postoperatively
  Grip strength was taken with a Jamar Dynamometer in the 2nd hand position.
Wrist Flexion | 10-14 days postoperatively
Lateral Pinch Strength | 10-14 days postoperatively
  Lateral pinch strength was taken with a Preston Pinch Gauge.

SECONDARY OUTCOMES:
Demographic Information | Preoperatively
  Sex, age, BMI, Smoking Status, Hand Dominance, Workers' Compensation Status
Complications | 10-14 days postoperatively
  Complications were observed for and recorded throughout the study.

OTHER OUTCOMES:
QuickDASH | 6 weeks postoperatively
  The Quick Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure was designed in 1998 with the goal of providing a more accurate depiction of the everyday symptoms and handicaps exclusively experienced by a patient with an upper extremity musculoskeletal condition. Designed as a patient-completed questionnaire, the DASH Outcome Measure can be administered multiple times throughout patient care to measure changes in function and symptoms over time
QuickDASH | 3 months postoperatively
  The Quick Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure was designed in 1998 with the goal of providing a more accurate depiction of the everyday symptoms and handicaps exclusively experienced by a patient with an upper extremity musculoskeletal condition. Designed as a patient-completed questionnaire, the DASH Outcome Measure can be administered multiple times throughout patient care to measure changes in function and symptoms over time
QuickDASH | 6 months postoperatively
  The Quick Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure was designed in 1998 with the goal of providing a more accurate depiction of the everyday symptoms and handicaps exclusively experienced by a patient with an upper extremity musculoskeletal condition. Designed as a patient-completed questionnaire, the DASH Outcome Measure can be administered multiple times throughout patient care to measure changes in function and symptoms over time
QuickDASH | 12 months postoperatively
  The Quick Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure was designed in 1998 with the goal of providing a more accurate depiction of the everyday symptoms and handicaps exclusively experienced by a patient with an upper extremity musculoskeletal condition. Designed as a patient-completed questionnaire, the DASH Outcome Measure can be administered multiple times throughout patient care to measure changes in function and symptoms over time
Levine-Katz Functional Status Scale (FSS) | 10-14 days postoperatively
  The Levine-Katz Functional Status Scale (FSS) has 8 questions self-rated on a 5-point scale on difficulty with 5 meaning so difficult patient is unable to perform the function.
Levine-Katz Functional Status Scale (FSS) | 6 weeks postoperatively
  The Levine-Katz Functional Status Scale (FSS) has 8 questions self-rated on a 5-point scale on difficulty with 5 meaning so difficult patient is unable to perform the function.
Levine-Katz Functional Status Scale (FSS) | 3 months postoperatively
  The Levine-Katz Functional Status Scale (FSS) has 8 questions self-rated on a 5-point scale on difficulty with 5 meaning so difficult patient is unable to perform the function.
Levine-Katz Functional Status Scale (FSS) | 6 months postoperatively
  The Levine-Katz Functional Status Scale (FSS) has 8 questions self-rated on a 5-point scale on difficulty with 5 meaning so difficult patient is unable to perform the function.
Levine-Katz Functional Status Scale (FSS) | 12 months postoperatively
  The Levine-Katz Functional Status Scale (FSS) has 8 questions self-rated on a 5-point scale on difficulty with 5 meaning so difficult patient is unable to perform the function.
Levine-Katz Symptom Severity Scale (SSS) | 6 weeks postoperatively
  The Levine-Katz Symptom Severity Scale (SSS) assesses pain, weakness, and sensation with 11 questions the patient rates on a 5-point scale with 5 indicating the most difficult; the average score is reported.
Levine-Katz Symptom Severity Scale (SSS) | 3 months postoperatively
  The Levine-Katz Symptom Severity Scale (SSS) assesses pain, weakness, and sensation with 11 questions the patient rates on a 5-point scale with 5 indicating the most difficult; the average score is reported.
Levine-Katz Symptom Severity Scale (SSS) | 6 months postoperatively
  The Levine-Katz Symptom Severity Scale (SSS) assesses pain, weakness, and sensation with 11 questions the patient rates on a 5-point scale with 5 indicating the most difficult; the average score is reported.
Levine-Katz Symptom Severity Scale (SSS) | 12 months postoperatively
  The Levine-Katz Symptom Severity Scale (SSS) assesses pain, weakness, and sensation with 11 questions the patient rates on a 5-point scale with 5 indicating the most difficult; the average score is reported.
Numerical Pain Rating Scale | 6 weeks postoperatively
  Patients are asked to describe their level of pain intensity over the last 24 hours. The pain scale anchor points 0 and 10 correspond to no pain and worst imaginable pain, respectively. The NPRS can be used multiple times throughout patient care, but has the greatest value in describing post-operative pain-related morbidity.
Numerical Pain Rating Scale | 3 months postoperatively
  Patients are asked to describe their level of pain intensity over the last 24 hours. The pain scale anchor points 0 and 10 correspond to no pain and worst imaginable pain, respectively. The NPRS can be used multiple times throughout patient care, but has the greatest value in describing post-operative pain-related morbidity.
Numerical Pain Rating Scale | 6 months postoperatively
  Patients are asked to describe their level of pain intensity over the last 24 hours. The pain scale anchor points 0 and 10 correspond to no pain and worst imaginable pain, respectively. The NPRS can be used multiple times throughout patient care, but has the greatest value in describing post-operative pain-related morbidity.
Numerical Pain Rating Scale | 12 months postoperatively
  Patients are asked to describe their level of pain intensity over the last 24 hours. The pain scale anchor points 0 and 10 correspond to no pain and worst imaginable pain, respectively. The NPRS can be used multiple times throughout patient care, but has the greatest value in describing post-operative pain-related morbidity.
Grip Strength | 6 weeks postoperatively
  Grip strength was taken with a Jamar Dynamometer in the 2nd hand position.
Grip Strength | 3 months postoperatively
  Grip strength was taken with a Jamar Dynamometer in the 2nd hand position.
Grip Strength | 6 months postoperatively
  Grip strength was taken with a Jamar Dynamometer in the 2nd hand position.
Grip Strength | 12 months postoperatively
  Grip strength was taken with a Jamar Dynamometer in the 2nd hand position.
Wrist Flexion | 6 weeks postoperatively
Wrist Flexion | 3 months postoperatively
Wrist Flexion | 6 months postoperatively
Wrist Flexion | 12 months postoperatively
Wrist Extension | 10-14 days postoperatively
Wrist Extension | 6 weeks postoperatively
Wrist Extension | 3 months postoperatively
Wrist Extension | 6 months postoperatively
Wrist Extension | 12 months postoperatively
Lateral Pinch Strength | 6 weeks postoperatively
  Lateral pinch strength was taken with a Preston Pinch Gauge.
Lateral Pinch Strength | 3 months postoperatively
  Lateral pinch strength was taken with a Preston Pinch Gauge.
Lateral Pinch Strength | 6 months postoperatively
  Lateral pinch strength was taken with a Preston Pinch Gauge.
Lateral Pinch Strength | 12 months postoperatively
  Lateral pinch strength was taken with a Preston Pinch Gauge.
Complications | 6 weeks postoperatively
  Complications were observed for and recorded throughout the study.
Complications | 3 months postoperatively
  Complications were observed for and recorded throughout the study.
Complications | 6 months postoperatively
  Complications were observed for and recorded throughout the study.
Complications | 12 months postoperatively
  Complications were observed for and recorded throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Bear, MD, Study Director — OrthoIllinois

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patterson JD, Simmons BP. Outcomes assessment in carpal tunnel syndrome. Hand Clin. 2002 May;18(2):359-63, viii. doi: 10.1016/s0749-0712(01)00002-6. PMID 12371039
- [Background] Jessurun W, Hillen B, Huffstadt AJ. Carpal tunnel release; postoperative care. Handchir Mikrochir Plast Chir. 1988 Jan;20(1):39-40. PMID 3350401
- [Background] Cook AC, Szabo RM, Birkholz SW, King EF. Early mobilization following carpal tunnel release. A prospective randomized study. J Hand Surg Br. 1995 Apr;20(2):228-30. doi: 10.1016/s0266-7681(05)80057-9. PMID 7797977
- [Background] Bhatia R, Field J, Grote J, Huma H. Does splintage help pain after carpal tunnel release? J Hand Surg Br. 2000 Apr;25(2):150. doi: 10.1054/jhsb.2000.0365. PMID 11062571
- [Background] Bury TF, Akelman E, Weiss AP. Prospective, randomized trial of splinting after carpal tunnel release. Ann Plast Surg. 1995 Jul;35(1):19-22. doi: 10.1097/00000637-199507000-00004. PMID 7574280
- [Background] Finsen V, Andersen K, Russwurm H. No advantage from splinting the wrist after open carpal tunnel release. A randomized study of 82 wrists. Acta Orthop Scand. 1999 Jun;70(3):288-92. doi: 10.3109/17453679908997810. PMID 10429608
- [Background] Martins RS, Siqueira MG, Simplicio H. Wrist immobilization after carpal tunnel release: a prospective study. Arq Neuropsiquiatr. 2006 Sep;64(3A):596-9. doi: 10.1590/s0004-282x2006000400013. PMID 17119800
- [Background] Ritting AW, Leger R, O'Malley MP, Mogielnicki H, Tucker R, Rodner CM. Duration of postoperative dressing after mini-open carpal tunnel release: a prospective, randomized trial. J Hand Surg Am. 2012 Jan;37(1):3-8. doi: 10.1016/j.jhsa.2011.10.011. Epub 2011 Nov 30. PMID 22133704
- [Background] Huisstede BM, Randsdorp MS, Coert JH, Glerum S, van Middelkoop M, Koes BW. Carpal tunnel syndrome. Part II: effectiveness of surgical treatments--a systematic review. Arch Phys Med Rehabil. 2010 Jul;91(7):1005-24. doi: 10.1016/j.apmr.2010.03.023. PMID 20599039
- [Background] Isaac SM, Okoro T, Danial I, Wildin C. Does wrist immobilization following open carpal tunnel release improve functional outcome? A literature review. Curr Rev Musculoskelet Med. 2010 Jul 11;3(1-4):11-7. doi: 10.1007/s12178-010-9060-9. PMID 21063494
- [Background] Keilani MY, Crevenna R, Fialka-Moser V. [Postoperative rehabilitation of patients with carpal tunnel syndrome]. Wien Med Wochenschr. 2002;152(17-18):479-80. doi: 10.1046/j.1563-258x.2002.01137.x. German. PMID 12385074
- [Background] Peters S, Page MJ, Coppieters MW, Ross M, Johnston V. Rehabilitation following carpal tunnel release. Cochrane Database Syst Rev. 2013 Jun 5;(6):CD004158. doi: 10.1002/14651858.CD004158.pub2. PMID 23740605
- [Background] Mathiowetz V, Weber K, Volland G, Kashman N. Reliability and validity of grip and pinch strength evaluations. J Hand Surg Am. 1984 Mar;9(2):222-6. doi: 10.1016/s0363-5023(84)80146-x. PMID 6715829
- [Background] Duncan KH, Lewis RC Jr, Foreman KA, Nordyke MD. Treatment of carpal tunnel syndrome by members of the American Society for Surgery of the Hand: results of a questionnaire. J Hand Surg Am. 1987 May;12(3):384-91. doi: 10.1016/s0363-5023(87)80011-4. PMID 3584886
- [Background] Leinberry CF, Rivlin M, Maltenfort M, Beredjiklian P, Matzon JL, Ilyas AM, Hutchinson DT. Treatment of carpal tunnel syndrome by members of the American Society for Surgery of the Hand: a 25-year perspective. J Hand Surg Am. 2012 Oct;37(10):1997-2003.e3. doi: 10.1016/j.jhsa.2012.07.016. PMID 23021173
- [Background] Shin EK, Bachoura A, Jacoby SM, Chen NC, Osterman AL. Treatment of carpal tunnel syndrome by members of the American Association for Hand Surgery. Hand (N Y). 2012 Dec;7(4):351-6. doi: 10.1007/s11552-012-9455-8. PMID 24294152
- [Background] Munns JJ, Awan HM. Trends in carpal tunnel surgery: an online survey of members of the American Society for Surgery of the Hand. J Hand Surg Am. 2015 Apr;40(4):767-71.e2. doi: 10.1016/j.jhsa.2014.12.046. Epub 2015 Mar 4. PMID 25747738
- [Result] Dziura JD, Post LA, Zhao Q, Fu Z, Peduzzi P. Strategies for dealing with missing data in clinical trials: from design to analysis. Yale J Biol Med. 2013 Sep 20;86(3):343-58. eCollection 2013 Sep. PMID 24058309